CLINICAL TRIAL: NCT00061828
Title: Childhood Liver Disease Research Network (ChiLDReN): A Prospective Database of Infants With Cholestasis
Brief Title: A Prospective Database of Infants With Cholestasis
Acronym: PROBE
Status: Recruiting | Type: Observational
Sponsor: Arbor Research Collaborative for Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: PROBE Study - ChiLDReN Network; U01DK103149 (NIH); U01DK103140 (NIH); U01DK103135 (NIH); U01DK084575 (NIH); U01DK084538 (NIH); U01DK084536 (NIH); U01DK062503 (NIH); U01DK062500 (NIH); U01DK062497 (NIH); U01DK062481 (NIH); U01DK062470 (NIH); U01DK062466 (NIH); U01DK062456 (NIH); U01DK062453 (NIH); U01DK062452 (NIH); U01DK062445 (NIH); U01DK062436 (NIH); U24DK062456 (NIH)
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Biliary Atresia
MeSH Terms: conditions — Biliary Atresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In this iteration of the study protocol only samples of blood will be collected for research purposes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Biliary Atresia: Infants presenting with cholestasis who are diagnosed with biliary atresia.

SUMMARY:
Biliary atresia, idiopathic neonatal hepatitis, and specific genetic cholestatic conditions are the most common causes of jaundice and hyperbilirubinemia that continue beyond the newborn period. The long term goal of the Childhood Liver Disease Research Network (ChiLDReN) is to establish a database of clinical information and plasma, serum, and tissue samples from cholestatic children to facilitate research and to perform clinical, epidemiological and therapeutic trials in these important pediatric liver diseases.

DETAILED DESCRIPTION:
This is a multi-center project to establish a prospective database of clinical information and a repository of blood, from children with diagnosis of neonatal liver disease, such as biliary atresia (BA), in order to perform research in this important liver problem. Children (diagnosed with BA or suspicious for BA) will be screened and enrolled at presentation at the participating pediatric liver sites. Participants diagnosed with BA will be followed intensively for the first year, at 18 months of age, and then annually up to 10 years of age, and then biannually, or liver transplantation. Other participants (Non-BA) diagnosed with cholestasis will be exited from the study at the time of diagnosis determination.

Detailed clinical data, laboratory investigations, liver and biliary specimens, and long-term follow-up of outcomes are part of the normal standard of care with respect to the diagnosis and treatment of the subjects with liver problems. This research involves the collection of diagnostic, clinical and outcome data concerning the subject, which is kept without identification (coded) in a national research database of infants with liver disease. Samples of blood will be obtained for later research analysis, whenever possible, at the time of clinically indicated blood draws or when there is IV access for a clinical procedure. All data from this study will be kept in a secure research database at the Scientific Data Coordinating Center (SDCC) and transferred to the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) data repository after the study ends.

ELIGIBILITY:
INCLUSION CRITERIA

* Infant's age less than or equal to 180 days at initial presentation at the ChiLDReN clinical site.
* Diagnosis of cholestasis defined by serum direct or conjugated bilirubin greater than or equal to 2 mg/dl and suspected biliary atresia.
* The subject's parent(s)/guardian(s) willing to provide informed written consent.

EXCLUSION CRITERIA

* Acute liver failure.
* Previous hepatobiliary surgery with dissection or excision of biliary tissue.
* Diagnoses of bacterial or fungal sepsis (except where associated with metabolic liver disease)
* Diagnoses of hypoxia, shock or ischemic hepatopathy within the past two weeks (If the cholestasis persists beyond two weeks of the initiating event, the infant can be enrolled).
* Diagnosis of any malignancy.
* Presence of any primary hemolytic disease (except when diagnosed with biliary atresia or another cholestatic disease being studied by ChiLDREN).
* Diagnosis of any drug or Total parenteral nutrition (TPN)-associated cholestasis (except when diagnosed with biliary atresia or another cholestatic disease being studied by ChiLDREN).
* Diagnosis with Extracorporeal membrane oxygenation (ECMO)-associated cholestasis.
* Birth weight less than 1500g (except when diagnosed with biliary atresia).

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study population will be selected from the patient base of participating specialty care clinics.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2004-04-21 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in disease severity over time (disease progression) | Measured at baseline, 1 month, 2 months, 3, 6 months post-baseline, 12 and 18 months of age, annually through year 10 and then biannually through year 20.
  disease progression defined by transplant date, date of death, worsening liver function, and complications related to worsening liver function

CONTACTS AND LOCATIONS:
Overall Officials: Saul Karpen, MD, PhD, Study Chair — VCU School of Medicine; Ed Doo, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); John Magee, MD, Principal Investigator — University of Michigan Medical Center, Ann Arbor; Lisa Henn, PhD, Principal Investigator — Arbor Research Collaborative for Health; Katrina Loh, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (16):
- United States (15):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta - Emory University, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The data will be transferred to NIDDK at the end of the study.

REFERENCES:
- [Derived] Teckman J, Rosenthal P, Ignacio RV, Spino C, Bass LM, Horslen S, Wang K, Magee JC, Karpen S, Asai A, Molleston JP, Squires RH, Kamath BM, Guthery SL, Loomes KM, Shneider BL, Sokol RJ; ChiLDReN (Childhood Liver Disease Research Network). Neonatal cholestasis in children with Alpha-1-AT deficiency is a risk for earlier severe liver disease with male predominance. Hepatol Commun. 2023 Dec 7;7(12):e0345. doi: 10.1097/HC9.0000000000000345. eCollection 2023 Dec 1. PMID 38055647
- [Derived] Kemme S, Canniff JD, Feldman AG, Garth KM, Li S, Pan Z, Sokol RJ, Weinberg A, Mack CL. Cytomegalovirus in biliary atresia is associated with increased pretransplant death, but not decreased native liver survival. Hepatol Commun. 2023 Jul 17;7(8):e0175. doi: 10.1097/HC9.0000000000000175. eCollection 2023 Aug 1. PMID 37471052
- [Derived] Hertel PM, Hawthorne K, Kim S, Finegold MJ, Shneider BL, Squires JE, Gupta NA, Bull LN, Murray KF, Kerkar N, Ng VL, Molleston JP, Bezerra JA, Loomes KM, Taylor SA, Schwarz KB, Turmelle YP, Rosenthal P, Magee JC, Sokol RJ; Childhood Liver Disease Research Network (ChiLDReN). Presentation and Outcomes of Infants With Idiopathic Cholestasis: A Multicenter Prospective Study. J Pediatr Gastroenterol Nutr. 2021 Oct 1;73(4):478-484. doi: 10.1097/MPG.0000000000003248. PMID 34310436
- [Derived] Ng VL, Sorensen LG, Alonso EM, Fredericks EM, Ye W, Moore J, Karpen SJ, Shneider BL, Molleston JP, Bezerra JA, Murray KF, Loomes KM, Rosenthal P, Squires RH, Wang K, Arnon R, Schwarz KB, Turmelle YP, Haber BH, Sherker AH, Magee JC, Sokol RJ; Childhood Liver Disease Research Network (ChiLDReN). Neurodevelopmental Outcome of Young Children with Biliary Atresia and Native Liver: Results from the ChiLDReN Study. J Pediatr. 2018 May;196:139-147.e3. doi: 10.1016/j.jpeds.2017.12.048. Epub 2018 Mar 5. PMID 29519540
- [Derived] Shneider BL, Magee JC, Karpen SJ, Rand EB, Narkewicz MR, Bass LM, Schwarz K, Whitington PF, Bezerra JA, Kerkar N, Haber B, Rosenthal P, Turmelle YP, Molleston JP, Murray KF, Ng VL, Wang KS, Romero R, Squires RH, Arnon R, Sherker AH, Moore J, Ye W, Sokol RJ; Childhood Liver Disease Research Network (ChiLDReN). Total Serum Bilirubin within 3 Months of Hepatoportoenterostomy Predicts Short-Term Outcomes in Biliary Atresia. J Pediatr. 2016 Mar;170:211-7.e1-2. doi: 10.1016/j.jpeds.2015.11.058. Epub 2015 Dec 24. PMID 26725209
- [Derived] Ye W, Rosenthal P, Magee JC, Whitington PF; Childhood Liver Disease Research and Education Network. Factors Determining delta-Bilirubin Levels in Infants With Biliary Atresia. J Pediatr Gastroenterol Nutr. 2015 May;60(5):659-63. doi: 10.1097/MPG.0000000000000690. PMID 25564820
- [Derived] Bessho K, Mourya R, Shivakumar P, Walters S, Magee JC, Rao M, Jegga AG, Bezerra JA. Gene expression signature for biliary atresia and a role for interleukin-8 in pathogenesis of experimental disease. Hepatology. 2014 Jul;60(1):211-23. doi: 10.1002/hep.27045. Epub 2014 May 27. PMID 24493287
- [Derived] Shneider BL, Abel B, Haber B, Karpen SJ, Magee JC, Romero R, Schwarz K, Bass LM, Kerkar N, Miethke AG, Rosenthal P, Turmelle Y, Robuck PR, Sokol RJ; Childhood Liver Disease Research and Education Network. Portal hypertension in children and young adults with biliary atresia. J Pediatr Gastroenterol Nutr. 2012 Nov;55(5):567-73. doi: 10.1097/MPG.0b013e31826eb0cf. PMID 22903006
- [Derived] Zahm AM, Hand NJ, Boateng LA, Friedman JR. Circulating microRNA is a biomarker of biliary atresia. J Pediatr Gastroenterol Nutr. 2012 Oct;55(4):366-9. doi: 10.1097/MPG.0b013e318264e648. PMID 22732895
- See also: Childhood Liver Disease Research Network (ChiLDReN) website — http://www.childrennetwork.org